CLINICAL TRIAL: NCT03382964
Title: A Randomized, Observer-Blinded, Dose-Escalation Phase 1 Study to Assess the Safety and Immunogenicity of Three Different Dose Levels of a Live-Attenuated Chikungunya Virus Vaccine Candidate (VLA1553) in Healthy Volunteers Aged 18 To 45 Years
Brief Title: Study to Assess the Safety and Immunogenicity of a Chikungunya Virus Vaccine Candidate (VLA1553) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA1553-101
Record Dates: First submitted 2017-12-12; First posted 2017-12-26 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Chikungunya
Keywords: VLA1553; Chikungunya; CHIKV; Live-attenuated Chikungunya virus vaccine
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VLA1553 low dose (Active Comparator): VLA1553 with 3.2x10^3 TCID50/ 100 µL (microliter). Re-vaccination at Month 12 with VLA1553 with 3.2x10^5 TCID50/ 1 mL (milliliter)
  Interventions: Biological: VLA1553
- VLA1553 medium dose (Active Comparator): VLA1553 with 3.2x10^4 TCID50/ 1 mL Re-vaccination at Month 12 with VLA1553 with 3.2x10^5 TCID50/ 1 mL
  Interventions: Biological: VLA1553
- VLA1553 high dose (Active Comparator): VLA1553 with 3.2x10^5 TCID50/ 1 mL Re-vaccination at Month 6 or Month 12 with VLA1553 with 3.2x10^5 TCID50/ 1 mL
  Interventions: Biological: VLA1553

INTERVENTIONS:
Biological: VLA1553 — I.M. vaccination with a live-attenuated Chikungunya virus (CHIKV) vaccine candidate

SUMMARY:
Randomized, observer-blinded, multicenter, dose-escalation Phase 1 clinical study investigating three dose levels of VLA1553 after a single immunization.

120 study participants will be enrolled into the study to receive three different doses (30 subjects in the low and medium and 60 subjects in the high dose group). Vaccination will be given intramuscularly on Day 0. As safety precaution, the study will begin with enrolment of 20 sentinel subjects in an open-label fashion. Thereafter, subjects will be enrolled in a blinded, randomized manner in the three study arms.

A re-vaccination will be given at Month 6 or Month 12 to confirm that a single vaccination will be sufficient to induce high titer neutralizing antibodies and protect subjects from CHIKV viremia.

Study participants will be followed up until 13 months after initial vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 45 years on the Day of screening;
* Has a BMI of ≥ 18.5 and < 30 kg/m2 on the Day of screening;
* Understanding of the study and its procedures, agrees to its provisions, and gives written informed consent prior to any study-related procedures;
* Generally healthy as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests;
* If female, subject is of non-childbearing potential. The definition of non-childbearing potential includes the following:

  1. Surgically sterile (e.g., hysterectomy with or without oophorectomy; fallopian tube ligation; endometrial ablation), at least 30 days prior to signature of the Informed Consent form;
  2. At least 5 years post-menopause (i.e., 6 years post last menstrual period), or menopause confirmed by follicle-stimulating hormone (FSH) testing.

Exclusion Criteria:

* History of known CHIKV infection;
* Plans to travel to areas with active CHIKV transmission during the course of the study or history of travel to an endemic CHIKV area within 4 weeks prior to study enrollment;
* Participation in a clinical study involving an investigational CHIKV vaccine;
* Receipt of an inactivated vaccine within 4 weeks or live vaccine within 8 weeks prior to vaccination in this study;
* Positive test results for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
* (1) Abnormal laboratory liver function values (≥ grade 1), (2) any grade 1 abnormal lab values deemed clinically relevant by the Investigator, and (3) any ≥ grade 2 abnormal lab values irrespective of clinical significance at screening;
* Clinically significant abnormal ECG at screening;
* History of significant cardiovascular, respiratory (including asthma), metabolic, neurological, hepatic, rheumatic, autoimmune, hematological, gastrointestinal or renal disorder;
* History of immune-mediated or clinically significant arthritis/arthralgia;
* History of malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved a cure;
* Disease or recent or current treatment that can be expected to influence immune response as specified in the protocol;
* History of severe hypersensitivity reactions or anaphylaxis;
* History of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications);
* Acute febrile infections within two weeks prior to vaccination;
* Subject is of childbearing potential or lactating at the time of enrollment;
* Blood donation within 30 days or receipt of blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or during the course of the study;
* A rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating;
* Known or suspected problem with alcohol or drug abuse as determined by the Investigator;
* Any condition that, in the opinion of the Investigator, may compromise the subjects well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
* Participation in another clinical study involving an investigational medicinal product within 30 days prior to study enrollment or during the course of this study;
* Member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2019-07-28 (Actual)

PRIMARY OUTCOMES:
Frequency of solicited injection site reactions | up to Day 14 after single vaccination
  Any measurable injection site reaction will be measured by size and includes injection site pain, tenderness, erythema/redness, induration and swelling.
Severity of solicited injection site reactions | up to Day 14 after single vaccination
  Any measurable injection site reaction will be measured by size and includes injection site pain, tenderness, erythema/redness, induration and swelling. They will be rated according to the Severity Grading Scale of Injection Site Reactions (FDA Guidance on Toxicity Grading Scales for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA 2007)
Frequency of solicited systemic reactions | up to Day 14 after single vaccination
  Systemic reactions including fever, nausea/vomiting, headache, fatigue, myalgia (muscle pain), arthralgia (joint pain) and rash will be reported in a standardized manner
Severity of solicited systemic reactions | up to Day 14 after single vaccination
  Systemic reactions including fever, nausea/vomiting, headache, fatigue, myalgia (muscle pain), arthralgia (joint pain) and rash will be reported in a standardized manner. They will be rated according to the FDA Guidance on Toxicity Grading Scales

SECONDARY OUTCOMES:
Frequency of any adverse event (AE) | until Day 14, Day 28 and throughout the study period
Severity of any adverse event (AE) | until Day 14, Day 28 and throughout the study period
  The investigator will assess the severity of AEs using his/her clinical expertise and judgment based on the most appropriate description (mild, moderate, severe) as per study protocol
Frequency of solicited injection site reactions | until Day 14, Day 28 and throughout the study period
  Any measurable injection site reaction will be measured by size and includes injection site pain, tenderness, erythema/redness, induration and swelling.
Severity of solicited injection site reactions | until Day 14, Day 28 and throughout the study period
  Any measurable injection site reaction will be measured by size and includes injection site pain, tenderness, erythema/redness, induration and swelling. They will be rated according to the Severity Grading Scale of Injection Site Reactions (FDA Guidance on Toxicity Grading Scales for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials (FDA 2007)
Frequency of solicited systemic reactions | until Day 14, Day 28 and throughout the study period
  Systemic reactions including fever, nausea/vomiting, headache, fatigue, myalgia (muscle pain), arthralgia (joint pain) and rash will be reported in a standardized manner
Severity of solicited systemic reactions | until Day 14, Day 28 and throughout the study period
  Systemic reactions including fever, nausea/vomiting, headache, fatigue, myalgia (muscle pain), arthralgia (joint pain) and rash will be reported in a standardized manner. They will be rated according to the FDA Guidance on Toxicity Grading Scales
Assessment of viremia after each vaccination | on Days 3, 7, 14 and beyond Day 14 after re-vaccination
  Assessment of CHIKV viremia will be done by RT (real-time)-qPCR (quantitative polymerase chain reaction) in blood and urine
Immune response as measured by CHIKV-specific neutralizing antibody titer as determined by micro-neutralization (μNT) assay. | Day 28, Day 84, Month 6, Month 12, and 28 days after re-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Nina Wressnigg, Study Chair — Valneva Austria GmbH
Locations (2):
- United States (2):
  - Optimal Research, LLC, Huntsville, Alabama
  - Optimal Research, LLC, Peoria, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wressnigg N, Hochreiter R, Zoihsl O, Fritzer A, Bezay N, Klingler A, Lingnau K, Schneider M, Lundberg U, Meinke A, Larcher-Senn J, Corbic-Ramljak I, Eder-Lingelbach S, Dubischar K, Bender W. Single-shot live-attenuated chikungunya vaccine in healthy adults: a phase 1, randomised controlled trial. Lancet Infect Dis. 2020 Oct;20(10):1193-1203. doi: 10.1016/S1473-3099(20)30238-3. Epub 2020 Jun 1. PMID 32497524